CLINICAL TRIAL: NCT03870542
Title: Multicenter, Prospective Observational Study to Identify and Validate a Composite of Urinary Exosomal Biomarkers for Kidney Allograft Tubulointerstitial Fibrosis
Brief Title: Multicenter, Prospective Study for Urinary Exosomal Biomarkers of Kidney Allograft Tubulointerstitial Fibrosis
Acronym: UFO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Korea University Anam Hospital (Other); Inje University (Other); Ulsan University Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Sung Shin, Associate Professor, Asan Medical Center
Other Study IDs: S2019-0362-0001
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Renal Fibrosis; Kidney Transplant Failure
MeSH Terms: interventions — Kidney Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine samples from deceased kidney donors, zero-day kidney graft biopsy specimen, Urine and blood samples of kidney transplant recipients during a follow up of one year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Deceased donor kidney transplantation: Patients receiving kidney transplants from deceased donor in the participating centers during the study period
  Interventions: Procedure: kidney transplantation

INTERVENTIONS:
Procedure: kidney transplantation — Kidney transplant for end-stage renal disease from deceased kidney donors

SUMMARY:
The investigators aim to identify urinary exosomal biomarkers that represent the extent of graft fibrosis from deceased donor kidney transplantation. Urinary samples will be collected from deceased kidney donors at the time of procurement and zero-day kidney graft biopsy will be performed at the time of transplant. The association between urinary exosomes and the degree of graft fibrosis will be analyzed to identify biomarkers that represent fibrosis. The correlation between these biomarkers and graft long term outcomes will be investigated.

DETAILED DESCRIPTION:
Interstitial fibrosis and tubular atrophy (IFTA), previously known as chronic allograft nephropathy (CAN), is diagnosed by pathologic changes involving all parts of the renal parenchyma and is one of the factors impacting graft survival and outcome. Currently, there is no standard to predict allograft fibrosis status at the time of procurement. Noninvasive biomarkers are necessary to monitor allograft status and to predict long-term outcomes.

The investigators aim to conduct a multicenter prospective study to identify urinary exosomal biomarkers that represent the extent of graft fibrosis from deceased donor kidney transplantation. Urinary samples will be collected from deceased kidney donors at the time of procurement and zero-day kidney graft biopsy will be performed at the time of transplant. The zero-day biopsy tissue will be stained with Masson's Trichrome staining, Collagen I, III, IV immunostaining to evaluate the degree of fibrosis. Also, by ultracentrifuge, we will extract urinary exosomes and perform proteomics analysis and RNA-sequencing. The association between urinary exosomes and the degree of graft fibrosis will be analyzed to identify biomarkers that represent fibrosis. The correlation between these biomarkers and graft long term outcomes will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* end-stage renal disease patients receiving kidney transplantation from deceased donors who have the ability to provide content for this study

Exclusion Criteria:

* multi-organ transplantation candidate or history of previous transplant, history of extra-renal solid organ or bone marrow or stem cell transplant, active infection, history of recent intoxication of alcohol or substance abuse within 24 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: end-stage renal disease patients receiving kidney transplantation from deceased donors who have the ability to provide content for this study, patients willing to provide content and participate in this study during the follow-up period
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-05-11 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
kidney fibrosis | zero-day (time of transplant)
  the degree of kidney graft fibrosis on zero day biopsy

SECONDARY OUTCOMES:
Kidney graft function | 6 months and 1 year post-transplant
  Kidney graft function assessed with serum Creatinine, eGFR, CKD-EPI

CONTACTS AND LOCATIONS:
Overall Officials: Sung Shin, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh T, Astor B, Zhong W, Mandelbrot D, Djamali A, Panzer S. Kidney Transplant Recipients With Primary Membranous Glomerulonephritis Have a Higher Risk of Acute Rejection Compared With Other Primary Glomerulonephritides. Transplant Direct. 2017 Oct 18;3(11):e223. doi: 10.1097/TXD.0000000000000736. eCollection 2017 Nov. PMID 29184911
- [Background] Hanssen O, Erpicum P, Lovinfosse P, Meunier P, Weekers L, Tshibanda L, Krzesinski JM, Hustinx R, Jouret F. Non-invasive approaches in the diagnosis of acute rejection in kidney transplant recipients. Part I. In vivo imaging methods. Clin Kidney J. 2017 Feb;10(1):97-105. doi: 10.1093/ckj/sfw062. Epub 2016 Jul 28. PMID 28643821
- [Background] Gamez-Valero A, Lozano-Ramos SI, Bancu I, Lauzurica-Valdemoros R, Borras FE. Urinary extracellular vesicles as source of biomarkers in kidney diseases. Front Immunol. 2015 Jan 30;6:6. doi: 10.3389/fimmu.2015.00006. eCollection 2015. PMID 25688242
- [Background] Li B, Hartono C, Ding R, Sharma VK, Ramaswamy R, Qian B, Serur D, Mouradian J, Schwartz JE, Suthanthiran M. Noninvasive diagnosis of renal-allograft rejection by measurement of messenger RNA for perforin and granzyme B in urine. N Engl J Med. 2001 Mar 29;344(13):947-54. doi: 10.1056/NEJM200103293441301. PMID 11274620
- [Background] Gonzalez-Nolasco B, Wang M, Prunevieille A, Benichou G. Emerging role of exosomes in allorecognition and allograft rejection. Curr Opin Organ Transplant. 2018 Feb;23(1):22-27. doi: 10.1097/MOT.0000000000000489. PMID 29189413